CLINICAL TRIAL: NCT05398367
Title: Effect of Single Ingredient and Blend Galactagogue Supplements on Increasing Milk Supply in Lactating Women Experiencing Diagnosed or Perceived Low Milk Supply
Brief Title: Galactagogue Use in Lactating Women With Low Milk Supply
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University (Other)
Responsible Party: Principal Investigator, Hope Lima, Assistant Professor and Graduate Director, Winthrop University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB22107R
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Breast Milk Expression
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of four treatment groups: Oat Mama Lactation Supplement (O), moringa supplement (M), shatavari supplement (S), or control (C).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Oat Mama Lactation Supplement (Experimental): Participants will receive a 20 day supply of oat mama lactation supplement for consumption per the manufacturer instructions
  Interventions: Dietary Supplement: Galactagogue Supplement for Treatment of Low Milk Supply
- Moringa Supplement (Experimental): Participants will receive a 20 day supply of moringa supplement for consumption per the manufacturer instructions
  Interventions: Dietary Supplement: Galactagogue Supplement for Treatment of Low Milk Supply
- Shatavari Supplement (Experimental): Participants will receive a 20 day supply of shatavari supplement for consumption per the manufacturer instructions
  Interventions: Dietary Supplement: Galactagogue Supplement for Treatment of Low Milk Supply
- Placebo (Placebo Comparator): Participants will receive a 20 day supply of placebo pills containing a mixture of flour and brown sugar. Participants will consume 2 placebo pills once per day for 20 days.
  Interventions: Dietary Supplement: Galactagogue Supplement for Treatment of Low Milk Supply

INTERVENTIONS:
Dietary Supplement: Galactagogue Supplement for Treatment of Low Milk Supply — Participants will consume a commercially available dietary supplement on the market for augmentation of breast milk production in lactating women with low milk supply

SUMMARY:
This study aims to determine whether a 20-day supplement with either Oat Mama Lactation Supplement, moringa, or shatavari has any impact on milk production through an increase in serum prolactin levels when compared to the placebo group. This data will be used to determine if clinical recommendations can be made for the use of the studied supplements in increasing milk supply.

DETAILED DESCRIPTION:
This study will be a double-blind randomized control trial where eligible participants will be randomized into one of four treatment groups: Oat Mama Lactation Supplement (O), moringa supplement (M), shatavari supplement (S), or control (C). All participants will receive a supplement or placebo for consumption throughout the 20-day trial period, and all participants will receive support from a lactation consultant once per week to receive appropriate guidance for increasing milk supply. 24-hour milk output will be recorded on day 1, 10, and 20 using either pre- and post-feeding weights, 24-hour pump output, or a combination of both. Additionally, blood samples will be taken on day 1, 10, and 20 and serum will be isolated for later analysis of serum prolactin levels.

ELIGIBILITY:
Inclusion Criteria: Participants in the study must:

* Be struggling with diagnosed or perceived low milk supply
* Be willing to consume a randomly assigned galactagogue or placebo supplement
* Be willing to provide a blood sample at each lactation consult (day 1, 10, 20)
* Be willing to provide 24-hour expressed milk volume either using pre- and post-feed weights, total pump output, or a combination of both on day 1, 10, and 20

Exclusion Criteria: Participants will be excluded if:

* They have a history of breast reduction
* They have a history of utilizing in vitro fertilization
* They are not a biological female with mammary glands present for producing milk
* They have consumed galactagogues with the intention of increasing their milk supply during the current lactation cycle
* They are under age 18 or above age 39

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Lactating women
Enrollment: 120 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Breast Milk Supply | Intervention will last 20 days and 24-hour breast milk expression volume will be measured on day 1, 10, and 20 and used to calculate change in 24-hour breast milk expression volume over the trial period
  Change in breast milk supply will be evaluated using 24-hour breast milk expression volume
Change in Serum Prolactin | Intervention will last 20 days and blood samples will be taken on day 1, 10, am 20 and change in serum prolactin will be measured using a human serum prolactin ELISA kit
  Change in serum prolactin levels will be evaluated by taking blood samples on day 1, 10, and 20 and measuring serum prolactin using a human serum prolactin ELISA kit

CONTACTS AND LOCATIONS:
Overall Officials: Hope K Lima, PhD, Principal Investigator — Winthrop University
Locations (1):
- Winthrop University, Rock Hill, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There will be no sharing of individual participant data to researchers outside of the experimental team.